CLINICAL TRIAL: NCT04390022
Title: Pilot Study to Evaluate the Potential of Ivermectin to Reduce COVID-19 Transmission
Brief Title: Sars-CoV-2/COVID-19 Ivermectin Navarra-ISGlobal Trial
Acronym: SAINT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Barcelona Institute for Global Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAINT
Record Dates: First submitted 2020-05-07; First posted 2020-05-15 (Actual); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Covid-19; Coronavirus Infection; SARS-CoV-2 Infection
Keywords: ivermectin
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: SAINT is a double-blind, randomized controlled trial with two parallel groups that evaluates the efficacy of ivermectin in reducing nasal viral carriage at seven days after treatment in SARS-CoV-2 infected patients who are at low risk of progression to severe disease.
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivermectin (Active Comparator): Participants on this arm will receive a single, oral dose of ivermectin 400 mcg/kg at the enrolment visit.
  Interventions: Drug: Ivermectin
- Placebo (Placebo Comparator): Participants on the arm will receive a single, oral dose of placebo tablets at the enrollment visit.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivermectin — Single dose of STROMECTOL® tablets at 400mcg/kg
  Other Names: Stromectol
  Arms: Ivermectin
Drug: Placebo — Placebo tablets will not match ivermectin but they will be administered by staff not involved in the clinical care.
  Arms: Placebo

SUMMARY:
SAINT is a double-blind, randomized controlled trial with two parallel groups that evaluates the efficacy of ivermectin in reducing nasal viral carriage at seven days after treatment in SARS-CoV-2 infected patients who are at low risk of progression to severe disease. The trial is currently planned at a single center in Navarra.

DETAILED DESCRIPTION:
SAINT is a double-blind, randomized controlled trial with two parallel groups that evaluates the efficacy of ivermectin in reducing nasal viral carriage at seven days after treatment in SARS-CoV-2 infected patients who are at low risk of progression to severe disease. The trial is currently planned at a single center in Navarra.

Participants will be randomized to receive a single dose of 400 mcg/kg ivermectin or a placebo. The randomization code will be generated by the trial statistician using blocks that ensure balance between the groups.

The allocation will be made by the investigator after obtaining informed consent, and confirmation of fulfillment of all inclusion and none of the exclusion criteria. The investigational product will be administered by a researcher not involved in patient care or participant follow up.

Participants will remain in the trial for a period of 28 days.

In the interests of public health and containing transmission of infection, trial visits will be conducted in the participant's home by a clinical trial team comprising nursing and medical members.

Subsequent visits will be to assess clinical and laboratory parameters.

A final study visit will be made for participants who withdraw prematurely from the study or are withdrawn by the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with COVID-19 in the emergency room of the Clínica Universidad de Navarra with a positive SARS-CoV-2 PCR.
2. Residents of the Pamplona basin ("Cuenca de Pamplona")
3. The patient should be aged 18 to 59 years
4. Negative pregnancy test for women of child bearing age*
5. The patient or his/her representative, have given consent to participate in the study.
6. The patient should, in the investigator's opinion, be able to comply with all the requirements of the clinical trial (including home follow up during isolation)

   * Women of child bearing age may participate if they use a safe contraceptive method for the entire period of the study and at least one month afterwards. A woman is considered to not have childbearing capacity if she is post-menopausal (minimum of 2 years without menstruation) or has undergone surgical sterilization (at least one month before the study)

Exclusion Criteria:

1. Known history of Ivermectin allergy
2. Hypersensitivity to any component of Stromectol®
3. COVID-19 Pneumonia

   * Diagnosed by the attending physician
   * Identified in a chest X-ray
4. Fever or cough present for more than 48 hours
5. Positive IgG against SARS-CoV-2 by rapid test
6. Age under 18 or over 60 years
7. The following co-morbidities (or any other disease that might interfere with the study in the eyes of the investigator):

   * Immunosuppression
   * Chronic Obstructive Pulmonary Disease
   * Diabetes
   * Hypertension
   * Obesity
   * Acute or chronic renal failure
   * History of coronary disease
   * History of cerebrovascular disease
   * Current neoplasm
8. Recent travel history to countries that are endemic for Loa loa (Angola, Cameroon, Central African Republic, Chad, Democratic Republic of Congo, Ethiopia, Equatorial, Guinea, Gabon, Republic of Congo, Nigeria and Sudan)
9. Current use of CYP 3A4 or P-gp inhibitor drugs such as quinidine, amiodarone, diltiazem, spironolactone, verapamil, clarithromycin, erythromycin, itraconazole, ketoconazole, cyclosporine, tacrolimus, indinavir, ritonavir or cobicistat. Use of critical CYP3A4 substrate drugs such as warfarin.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2020-09-17 (Actual); Study Completion 2020-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos J Chaccour, MD PhD, Principal Investigator — Clinica Universidad de Navarra and Barcelona Institute of Global Health
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Navarre, Spain

REFERENCES:
- [Derived] Chaccour C, Casellas A, Blanco-Di Matteo A, Pineda I, Fernandez-Montero A, Ruiz-Castillo P, Richardson MA, Rodriguez-Mateos M, Jordan-Iborra C, Brew J, Carmona-Torre F, Giraldez M, Laso E, Gabaldon-Figueira JC, Dobano C, Moncunill G, Yuste JR, Del Pozo JL, Rabinovich NR, Schoning V, Hammann F, Reina G, Sadaba B, Fernandez-Alonso M. The effect of early treatment with ivermectin on viral load, symptoms and humoral response in patients with non-severe COVID-19: A pilot, double-blind, placebo-controlled, randomized clinical trial. EClinicalMedicine. 2021 Feb;32:100720. doi: 10.1016/j.eclinm.2020.100720. Epub 2021 Jan 19. PMID 33495752

RESULTS

PARTICIPANT FLOW:
Groups:
- Ivermectin: Participants on this arm received a single, oral dose of ivermectin 400 mcg/kg at the enrolment visit.
  (Single dose of STROMECTOL® tablets at 400mcg/kg)
- Placebo: Participants on this arm received a single, oral dose of placebo tablets at the enrollment visit.
  (Placebo tablets did not match ivermectin but they were administered by staff not involved in the clinical care)
Period: Overall Study
Arm/Group | Ivermectin | Placebo
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ivermectin | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26 [19 to 36] | 26 [21 to 44] | 26 [20 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 7 | 5 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 23.5 [19.6 to 27.8] | 22.9 [21.0 to 24.8] | 22.9 [20.6 to 26.1]
Any symptoms [Count of Participants; unit: Participants] | 12 | 12 | 24
Earliest start of any symptom [Median (Inter-Quartile Range); unit: hours] — Presence of symptoms as well as their onset date was self-reported by each patient in the baseline visit.
  hours | 24 [24 to 48] | 48 [36 to 48] | 48 [24 to 48]
Fever [Count of Participants; unit: Participants] | 7 | 9 | 16
Earliest start of fever [Median (Inter-Quartile Range); unit: hours] — Presence of fever as well as its onset date was self-reported by each patient in the baseline visit. Population: Only patients with reported fever
  hours
    number analyzed (Participants) | 7 | 9 | 16
    (all) | 24 [12 to 24] | 24 [24 to 48] | 24 [15 to 36]
Cough [Count of Participants; unit: Participants] | 4 | 2 | 6
Earliest start of cough [Median (Inter-Quartile Range); unit: hours] — Presence of cough as well as its onset date was self-reported by each patient in the baseline visit. Population: Only patients with cough.
  hours
    number analyzed (Participants) | 4 | 2 | 6
    (all) | 24 [16 to 36] | 10 [8 to 12] | 18 [8 to 24]
CRP [Median (Inter-Quartile Range); unit: mg/dL] | 0.3 [0.2 to 0.8] | 0.3 [0.2 to 0.6] | 0.3 [0.2 to 0.7]
Ferritin [Median (Inter-Quartile Range); unit: mg/dL] | 165.0 [95.8 to 241.3] | 156.1 [103.1 to 223.0] | 160.9 [101.8 to 223.0]
IL-6 [Median (Inter-Quartile Range); unit: pg/mL] | 6.5 [5.1 to 9.6] | 4.5 [3.0 to 6.5] | 5.3 [3.8 to 8.2]
D-Dimer [Median (Inter-Quartile Range); unit: ng/mL] | 295 [270 to 420] | 280 [270 to 315] | 285 [270 to 365]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With a Positive SARS-CoV-2 PCR
Description: Proportion of patients with a positive SARS-CoV-2 PCR from a nasopharyngeal swab at day 7 post-treatment. PCRs were performed using two target genes (E and N).
Time Frame: 7 days post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Ivermectin | Placebo
Number analyzed (Participants) | 12 | 12
Participants
  PCR positivity (gene N) | 12 | 12
  PCR positivity (gene E) | 11 | 12

2. Secondary Outcome: Median Viral Load
Description: Quantitative and semi-quantitative PCR in nasopharyngeal swab. PCRs were performed using two target genes (E and N).
Time Frame: Baseline and on days 4, 7, 14 and 21
Measure: Median (Inter-Quartile Range); unit: copies/mL
Arm/Group | Ivermectin | Placebo
Number analyzed (Participants) | 12 | 12
copies/mL
  Gene E - day 1 | 16850000 [5915000 to 385250000] | 26700000 [8325000 to 423500000]
  Gene E - day 4 | 161000 [2820 to 878000] | 493500 [103700 to 9910000]
  Gene E - day 7 | 1018 [92 to 15445] | 23550 [709 to 226500]
  Gene E - day 14 | 7 [0 to 42] | 30 [1 to 50]
  Gene E - day 21 | 1 [0 to 9] | 0 [0 to 16]
  Gene N - day 1 | 367000000 [18350000 to 9280000000] | 327500000 [58300000 to 6740000000]
  Gene N - day 4 | 269000 [1885 to 1046500] | 2194500 [73150 to 37100000]
  Gene N - day 7 | 2255 [938 to 34650] | 36800 [4510 to 630500]
  Gene N - day 14 | 86 [0 to 1235] | 75 [24 to 710]
  Gene N - day 21 | 0 [0 to 67] | 107 [0 to 183]

3. Secondary Outcome: Fever and Cough Progression
Description: Proportion of patients with fever and cough
Time Frame: Days 4, 7, 14 and 21
Measure: Count of Participants; unit: Participants
Arm/Group | Ivermectin | Placebo
Number analyzed (Participants) | 12 | 12
Participants
  Fever - Day 4 | 0 | 0
  Fever - Day 7 | 1 | 0
  Fever - Day 14 | 0 | 0
  Fever - Day 21 | 0 | 0
  Cough - Day 4 | 5 | 6
  Cough - Day 7 | 5 | 5
  Cough - Day 14 | 1 | 3
  Cough - Day 21 | 1 | 3

4. Secondary Outcome: Seroconversion at Day 21
Description: Proportion of participants with positive IgG at day 21
Time Frame: Up to and including day 21
Measure: Count of Participants; unit: Participants
Arm/Group | Ivermectin | Placebo
Number analyzed (Participants) | 12 | 12
Participants | 12 | 12

5. Secondary Outcome: Proportion of Drug-related Adverse Events
Description: Proportion of drug-related adverse events
Time Frame: 7 days post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Ivermectin | Placebo
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

6. Secondary Outcome: Levels of IgG, IgM and IgA
Description: Levels in median fluorescence intensity (MFI) of IgG, IgM and IgA against the receptor-binding domain of the spike glycoprotein of SARS-CoV-2 in plasma, measured by a Luminex assay.
  [Results not yet available]
Time Frame: Up to and including day 28
Reporting Status: Not Posted

7. Secondary Outcome: Frequency of Innate Immune Cells
Description: Frequency (% over total PBMC) of innate immune cells (myeloid and plasmacytoid dendritic cells, NK cell, classical, intermediate and pro-inflammatory macrophages) measured in cryopreserved PBMC by flow cytometry.
  [Results not yet available]
Time Frame: Up to and including day 7
Reporting Status: Not Posted

8. Secondary Outcome: Frequency SARS-CoV-2-specific CD4+ T and and CD8+ T Cells
Description: Frequency of CD4+ T and CD8+ T cells (% over total CD4+T and CD8+ T) expressing any functional marker upon in vitro stimulation of PBMC with SARS-CoV-2 peptides, measured by flow cytometry.
  [Results not yet available]
Time Frame: Up to and including day 7
Reporting Status: Not Posted

9. Secondary Outcome: Results From Cytokine Human Magnetic 30-Plex Panel
Description: Concentration (all in pg/mL) of epidermal growth factor (EGF), fibroblast growth factor (FGF), granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), hepatocyte growth factor (HGF), vascular endothelial growth factor (VEGF), tumour necrosis factor (TNF), interferon (IFN)-α, IFN-γ, interleukin (IL)-1RA, IL-1β, IL-2, IL-2R, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12(p40/p70), IL-13, IL-15, IL-17, IFN-γ induced protein (IP-10), monocyte chemoattractant protein (MCP-1), monokine induced by IFN-γ (MIG), macrophage inflammatory protein (MIP)-1α, MIP-1β in plasma measured by a Luminex assay using a commercially available kit (Cytokine Human Magnetic 30-Plex Panel from ThermoFisher).
  [Results not yet available]
Time Frame: Up to and including day 28
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 28 days
Description: Adverse events were assessed at each study visit (days 1, 4, 7, 14, 21 and 28)
Arm/Group | Ivermectin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/12 | 5/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivermectin (N=12) | Placebo (N=12)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Insomnia (Nervous system disorders) | 0 (0) | 1 (1)
Ferritin elevation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute pharyngitis (tonsillitis) (Infections and infestations) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Hypochromic Microcytic Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dorsal discomfort of a mechanical nature (Cardiac disorders) | 1 (1) | 0 (0)
Worsening of acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abdominal bacterial translocation (Infections and infestations) | 0 (0) | 1 (1)
Hematoma (General disorders) | 1 (1) | 1 (1)
D-Dimer increase (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cold Sore (Cardiac disorders) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Grade II burn (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT04390022/SAP_000.pdf
  • Study Protocol (2020-08-12): https://cdn.clinicaltrials.gov/large-docs/22/NCT04390022/Prot_001.pdf